CLINICAL TRIAL: NCT06447090
Title: Study on the Efficacy and Safety of VMAC Combined With Donor Lymphocyte Infusion (DLI) in the Treatment of Patients With Relapse of Acute Myeloid Leukemia After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: VMAC+DLI Treatment of Patients With Relapse of AML After Allo-HSCT
Acronym: VMAC+DLI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024002
Record Dates: First submitted 2024-06-03; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Relapse Acute Myeloid Leukemia
Keywords: Mitoxantrone liposome
MeSH Terms: interventions — venetoclax; Cytarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VMAC+DLI (Experimental): VMAC regimen :
  Veneclatra (VEN) 400 mg/d (reduced to 100 mg when combined with an azole), d1-7; Mitoxantrone Liposomal 30 mg/m2, d1; Cytosine arabinoside(Ara-C) 100 mg/m2/d, d1-7; Cyclophosphamide (CTX) 400 mg/m2/d, d2, 5); After 1 day of rest, cryopreserved donor stem cells MNC1-2X10^8 /kg infusion, add low-dose (25 mg Bid) and short-course treatment (stop 2-3 weeks after DLI) oral cyclosporine (CSA) to prevent graft-versus-host disease (GVHD) 3 days before cryopreserved stem cell infusion.
  Interventions: Drug: Mitoxantrone hydrochloride liposome

INTERVENTIONS:
Drug: Mitoxantrone hydrochloride liposome — Veneclatra (VEN) 400 mg/d (reduced to 100 mg when combined with an azole), d1-7; Mitoxantrone Liposomal 30 mg/m2, d1; Cytosine arabinoside(Ara-C) 100 mg/m2/d, d1-7; Cyclophosphamide (CTX) 400 mg/m2/d, d2, 5); After 1 day of rest, cryopreserved donor stem cells MNC1-2X10^8 /kg infusion, add low-dose (25 mg Bid) and short-course treatment (stop 2-3 weeks after DLI) oral cyclosporine (CSA) to prevent graft-versus-host disease (GVHD) 3 days before cryopreserved stem cell infusion.
  Other Names: Venetoclax; Cytarabine,Cytosine arabinoside; Cyclophosphamide

SUMMARY:
This clinical trial included 30 cases and aimed to understand the effectiveness and safety of the VMAC regimen combined with donor lymphocyte infusion (DLI) in the treatment of patients with acute myeloid leukemia who have relapsed after allogeneic hematopoietic stem cell transplantation.

The main questions it aims to answer are:

The safety and efficacy of VMAC combined with DLI in the treatment of allo HSCT recurrence in AML patients;

DETAILED DESCRIPTION:
venetoclax 400 mg/d (reduced to 100 mg when combined with an azole), d1-7; liposomal mitoxantrone 30 mg/m2/d, d1; cytarabine (Ara-C) 100 mg/m2/d, d1-7; cyclophosphamide (CY) 400 mg/m2/d, d2, 5)，and then rest for 1 day before giving cryopreserved donor stem cells.MNC1-2X10^8/kg infusion, low-dose (25 mg Bid), short-course treatment (2-3 weeks after DLI) oral cyclosporine (CSA) is added to prevent graft-versus-host disease starting 3 days before the infusion of cryopreserved stem cells.

Monitor the occurrence of serious infections, cardiac toxicity, GVHD and other adverse reactions during the medication process; Blood routine recovery or bone marrow re examination 4 weeks after DLI to evaluate the efficacy of one course of VMAC combined with DLI; The patient was followed up for 2 years to evaluate long-term efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AML confirmed by bone marrow morphology and morphological recurrence after allo-HSCT (proportion of bone marrow morphological blast cells ≥5%);
2. Age ≥18 years and ≤65 years old, regardless of gender;
3. Eastern Oncology The evaluation of physical status of the cooperative group (ECOG-PS) is 0-2 points;
4. An informed consent form must be signed before the start of the research procedure, and the patient himself or his immediate family members must sign the informed consent form. Considering the patient's condition, if the patient's signature is not conducive to the treatment of the condition, the legal guardian or the patient's immediate family member will sign the informed consent form.

Exclusion Criteria:

Subjects who meet any of the following criteria shall not be enrolled in this study:

* 1) Secondary transplant patients;
* 2) Have a history of tumor and have received any treatment for this tumor in the past 3 years, except for superficial bladder cancer , basal cell or squamous cell carcinoma of the skin, cervical intraepithelial carcinoma (CIN) or prostate intraepithelial carcinoma (PIN);
* 3) Serological reactions of known HIV, active hepatitis B, and active hepatitis C virus positive or syphilis positive;
* 4) Suffering from mental illness or other conditions and unable to cooperate with the requirements of research treatment and monitoring;
* 5) Pregnant patients or patients who cannot take appropriate contraceptive measures during treatment;
* 6) Active heart disease, definition One or more of the following:

  1. Long QTc syndrome or QTc interval >480ms;
  2. Complete left bundle branch block, II or III degree atrioventricular block;
  3. Need for drug treatment or History of severe arrhythmia with clinical symptoms;
  4. New York Heart Association classification ≥ II;
  5. Left ventricular ejection fraction less than 50%;
  6. Myocardial infarction, unstable angina, severe myocardial infarction within 6 months before enrollment History of unstable ventricular arrhythmias or any other arrhythmias requiring treatment, clinically severe pericardial disease, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* 7) Transplantation from an unrelated donor;
* 8) Those deemed not suitable for enrollment by the researcher.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
CRR | 1 year
  All tumor target lesions disappear, no new lesions appear, and tumor markers are normal, maintained for at least 4 weeks

SECONDARY OUTCOMES:
PR | 1 year
  The maximum sum of diameters of tumor lesions decrease≥ 30% and is maintained for at least 4 weeks
ORR | 1year
  CR+PR
2-year OS | 2 years
  The time from the start of treatment to death due to any reason
DFS | 2 years
  The time from the start of treatment to disease recurrence or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Xin Chen, Doctor, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, China, Tianjin, Tianjin Municipality, China